CLINICAL TRIAL: NCT05645536
Title: Open-label, Safety Extension Study for Subjects With HR+, HER2-Negative Breast Cancer Who Have Completed the OVarian Suppression Evaluating Subcutaneous LeuprolIde Acetate in Breast Cancer OVELIA Study
Brief Title: Safety Extension Study for Subjects With HR+, HER2- Breast Cancer for Subjects Who Have Completed the OVELIA Study
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Tolmar Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOL2506A-EXT
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: Ovarian Suppression; HR+; HER2-; Oncology; Premenopausal
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Tamoxifen; Letrozole; Anastrozole; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TOL2506 (Experimental): TOL2506 in combination with standard endocrine therapy (Tamoxifen & Aromatase Inhibitors)
  Interventions: Drug: TOL2506; Drug: Tamoxifen; Drug: Letrozole tablets; Drug: Anastrozole Tablets; Drug: Exemestane Tablets

INTERVENTIONS:
Drug: TOL2506 — Leuprolide Acetate for injectable suspension, 30 mg. Subcutaneous injection every 3 months
Drug: Tamoxifen — 20 mg once daily or 10 mg 2 times daily - either tablet of solution
Drug: Letrozole tablets — One 2.5 mg tablet taken orally once daily
Drug: Anastrozole Tablets — One 1 mg tablet taken orally once daily
Drug: Exemestane Tablets — One 25 mg tablet taken orally once daily

SUMMARY:
TOL2506A (OVELIA) is a Phase 3, single arm, open-label study evaluating the effectiveness of TOL2506 in suppressing ovarian function in premenopausal women with HR+, HER2-negative breast cancer and men with HR+ breast cancer. The TOL2506A-EXT study described here is a safety extension study to assess and collect long-term data on the ongoing safety and tolerability of TOL2506 in combination with tamoxifen or an AI for up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

Females:

1. Completed Visit 9, Week 48 visit of TOL2506A study and is a candidate for continued endocrine therapy + ovarian suppression
2. Able to understand the investigational nature of this study and provide written informed consent prior to the participation in the trial
3. Age 18 to 51 inclusive

Exclusion Criteria:

* Females:

  1. Body mass index (BMI) < 18.00 kg/m2
  2. Life expectancy < 12 months
  3. ECOG performance status ≥ 3
  4. Unacceptable hepatic function as determined by any of the following:

     1. Alanine aminotransferase (ALT) ≥ 2X upper limit of normal (ULN)
     2. Aspartate aminotransferase (AST) ≥ 2X ULN
     3. Bilirubin ≥ 2X ULN
     4. Alkaline phosphatase ≥ 2X ULN
     5. Severe hepatic impairment (Child-Pugh Class C)
  5. Unacceptable renal function as determined by any of the following:

     1. Creatinine ≥ 3X ULN
     2. Creatinine clearance ≤ 30 mL/minute
     3. Creatinine clearance ≤ 60 mL/minute in subjects with bone density 1.5 standard deviations below the young adult normal mean
  6. Screening 12-lead ECG demonstrating any of the following:

     1. Heart rate > 100 beats per minute (BPM)
     2. QRS > 120 msec
     3. Corrected QT (QTc) > 450 msec
     4. PR > 220 msec
  7. Use of any new medications known to prolong the QT/QTc interval
  8. Any new medical condition or psychiatric, addictive or other disorder that, in the opinion of the Investigator, may interfere with trial conduct or result in the subject being ineligible to continue treatment with TOL2506
  9. Concomitant use of medications that may impact subject safety including but not limited to:

     1. Oral or transdermal hormonal therapy
     2. Estrogen, progesterone, or androgens
     3. Hormonal contraceptives
  10. Change in tolerability to TOL2506 that precludes continued treatment
  11. Sexually active with a male partner and not willing to use at least 2 non-hormonal contraceptive methods throughout the study
  12. Is of childbearing potential with a positive urine pregnancy test at Screening

Males:

Inclusion Criteria:

1. Completed Visit 9, Week 48 visit of TOL2506A study and is a candidate for continued endocrine + GnRH agonist therapy
2. Able to understand the investigational nature of this study and provide written informed consent prior to participation in the trial

Males:

Exclusion Criteria:

1. BMI < 18.00 kg/m2
2. Life expectancy < 12 months
3. ECOG performance status ≥ 3
4. Unacceptable hepatic function as determined by any of the following:

   1. ALT ≥ 2X ULN
   2. AST ≥ 2X ULN
   3. Bilirubin ≥ 2X ULN
   4. Alkaline phosphatase ≥ 2X ULN
   5. Severe hepatic impairment (Child-Pugh Class C)
5. Unacceptable renal function as determined by any of the following:

   1. Creatinine ≥ 3X ULN
   2. Creatinine clearance ≤ 30 mL/minute
   3. Creatinine clearance ≤ 60 mL/minute in subjects with bone density 1.5 standard deviations below the young adult normal mean
6. Screening 12-lead ECG demonstrating any of the following:

   1. HR > 100 BPM
   2. QRS > 120 msec
   3. QTc > 450 msec
   4. PR > 220 msec
7. Use of any new medications known to prolong the QT/QTc interval
8. Any new medical condition or psychiatric, addictive or other disorder that, in the opinion of the Investigator, may interfere with trial conduct or result in the subject being ineligible to continue treatment with TOL2506
9. Concomitant use of medications that may impact subject safety including but not limited to oral or transdermal hormonal therapy
10. Change in tolerability to TOL2506 that precludes continued treatment.

Ages: 18 Years to 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
The occurrences of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | 4 years from enrolling in study

CONTACTS AND LOCATIONS:
Locations (47):
- United States (17):
  - Marin Cancer Care, Inc., Greenbrae, California
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Baptist Health Lexington, Lexington, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Hematology Oncology Associates of Central New York, PC, East Syracuse, New York
  - Cape Fear Valley Health Systems - Cancer Center, Fayetteville, North Carolina
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Tennessee Oncology, PLLC, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology - Central South, Austin, Texas
  - Texas Oncology - Presbyterian Cancer Center, Dallas, Texas
  - Texas Oncology - Northeast Texas, Longview, Texas
  - Joe Arrington Cancer Research and Treatment Center at Covenant Children's Hospital, Lubbock, Texas
  - Texas Oncology - San Antonio, New Braunfels, Texas
  - Texas Oncology - DFW, Plano, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Argentina (6):
  - Instituto Medico de la Fundacion Estudios Clinicos, Rosario, Santa Fe Province
  - Hospital Aleman, Caba
  - Fundacion CENIT, CABA
  - Instituto Oncologico de Cordoba (IONC), Córdoba
  - Centro Privado de MRI de Rio Cuarto SA, Córdoba
  - Sanatorio Allende, Córdoba
- Brazil (9):
  - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Hospital Araujo Jorge, Goiânia, Goiás
  - Hospital do Cancer de Londrina, Londrina, Paraná
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Uniao Brasileira de Educacao e Assistencia, Porto Alegre, Rio Grande do Sul
  - Hospital de Amor Amazonia, Porto Velho, Rondônia
  - Instituto de Educacao, Pesquisa e Gestao em Saude, Rio de Janeiro
  - Centro de Estudos e Pesquisa de Hematologia e Oncologia, Santo André
  - Fundacao Pio XII - Hospital de Amor Barretos, São Paulo
- India (9):
  - Unique Hospital Multispecialty & Research Institute, Surat, Gujarat
  - SRV AGADI Hospital and Research Centre, Bangalore, Karnataka
  - Oncoville Cancer Hospital and Research Centre, Bengaluru, Karnataka
  - Mysore Medical College and Research Institute, Mysore, Karnataka
  - KIMS - Kingsway Hospitals, Nagpur, Maharashtra
  - HCG Manavata Cancer Centre, Nashik, Maharashtra
  - Indrayani Hospital and Cancer Institute, Pune, Maharashtra
  - Erode Cancer Centre Private Ltd., Erode, Tamil Nadu
  - Swami Harshankaranand Ji Hospital & Research Centre, Varanasi, Uttar Pradesh
- Mexico (5):
  - Unidad de Medicina Especializada SMA, San Juan del Río, Querétaro
  - CIMET Scientific Corporation S. A. P. I. de C. V., Guadalajara
  - Amiisto Atencion Medica Integral, Investigacion Y Terapia Oncologica S. A. DE C. V., Madero
  - Atencion Medica Integral E Investigacion en Terapia Oncologica, Mexico City
  - Faicic S de Rl de C. V., Veracruz
- FDI Clinical Research, San Juan, Puerto Rico